CLINICAL TRIAL: NCT01658501
Title: Phase 2b Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group Study to Assess the Pharmacodynamic Response and Safety of Three Dose Levels of (PB1023) Injection Following 20 Weeks of Once-Weekly Subcutaneous Dosing in Adult Subjects With Inadequately Treated Type 2 Diabetes Mellitus
Brief Title: Phase 2b Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group Study to Assess the PD Response and Safety of Three Dose Levels of (PB1023) Injection Following 20 Weeks of Weekly SC Dosing in Adults With T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB1023-PT-CL-0004
Record Dates: First submitted 2012-07-24; First posted 2012-08-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride; Liraglutide; Diet; Exercise; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Diet and Exercise (Experimental): Diet and exercise only.
  Interventions: Drug: 50 mg PB1023; Drug: 70 mg PB1023; Drug: 100 mg PB1023; Drug: Placebo (0.9% Sodium Chloride); Drug: Victoza®
- Metformin (Experimental): Metformin only
  Interventions: Drug: 50 mg PB1023; Drug: 70 mg PB1023; Drug: 100 mg PB1023; Drug: Placebo (0.9% Sodium Chloride); Drug: Victoza®
- Sulfonylurea (Experimental): Sulfonylurea only
  Interventions: Drug: 50 mg PB1023; Drug: 70 mg PB1023; Drug: 100 mg PB1023; Drug: Placebo (0.9% Sodium Chloride); Drug: Victoza®
- Metformin and Sulfonylurea (Experimental): Metformin and Sulfonylurea combination therapy
  Interventions: Drug: 50 mg PB1023; Drug: 70 mg PB1023; Drug: 100 mg PB1023; Drug: Placebo (0.9% Sodium Chloride); Drug: Victoza®
- PB1023 (Experimental): PB1023 weekly SC injection
  Interventions: Drug: 50 mg PB1023; Drug: 70 mg PB1023; Drug: 100 mg PB1023; Other: Diet and Exercise; Drug: Metformin; Drug: Sulfonylurea; Drug: Metformin and Sulfonylurea
- Placebo Comparator (Placebo Comparator): Placebo (0.9% Sodium Chloride) weekly SC injection
  Interventions: Drug: Placebo (0.9% Sodium Chloride); Other: Diet and Exercise; Drug: Metformin; Drug: Sulfonylurea; Drug: Metformin and Sulfonylurea
- Active Comparator (Active Comparator): Active Comparator (Victoza) daily SC injection
  Interventions: Drug: Victoza®; Other: Diet and Exercise; Drug: Metformin; Drug: Sulfonylurea; Drug: Metformin and Sulfonylurea

INTERVENTIONS:
Drug: 50 mg PB1023
  Arms: Diet and Exercise; Metformin; Metformin and Sulfonylurea; PB1023; Sulfonylurea
Drug: 70 mg PB1023
  Arms: Diet and Exercise; Metformin; Metformin and Sulfonylurea; PB1023; Sulfonylurea
Drug: 100 mg PB1023
  Arms: Diet and Exercise; Metformin; Metformin and Sulfonylurea; PB1023; Sulfonylurea
Drug: Placebo (0.9% Sodium Chloride)
  Other Names: SC Weekly Injection
  Arms: Diet and Exercise; Metformin; Metformin and Sulfonylurea; Placebo Comparator; Sulfonylurea
Drug: Victoza®
  Other Names: daily SC injection
  Arms: Active Comparator; Diet and Exercise; Metformin; Metformin and Sulfonylurea; Sulfonylurea
Other: Diet and Exercise
  Arms: Active Comparator; PB1023; Placebo Comparator
Drug: Metformin
  Arms: Active Comparator; PB1023; Placebo Comparator
Drug: Sulfonylurea
  Arms: Active Comparator; PB1023; Placebo Comparator
Drug: Metformin and Sulfonylurea
  Arms: Active Comparator; PB1023; Placebo Comparator

SUMMARY:
Primary objective:

The primary objective of this study is to define the dose response of Glymera as measured as the change from baseline in hemoglobin A1c (HbA1c) following 20 weeks of once-weekly dosing.

Secondary objectives:

The secondary objectives are to:

* Describe incidence, severity, and duration of reported gastrointestinal side effects of Glymera compared to active comparator;
* Compare change from baseline in HbA1c following 20 weeks of dosing compared to placebo and active comparator;
* Compare change from baseline in fasting plasma glucose (FPG) following 20 weeks of dosing compared to placebo and active comparator;
* Describe the frequencies of adverse events in the treatment groups; and
* Describe the above endpoints for the following subgroups of subjects according to baseline type 2 diabetes mellitus (T2DM) therapy: diet and exercise only, metformin only, sulfonylurea only, or metformin and sulfonylurea combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 75 years of age, inclusive;
* Body mass index ≤45 kg/m2;
* Diagnosed with T2DM with HbA1c of ≥7.0% and ≤11.0% and treated with diet and exercise alone, or with stable doses of metformin alone, sulfonylurea alone or metformin and sulfonylurea.

Exclusion Criteria:

* Currently taking or have taken within the last 6 months non-oral antihyperglycemic agents (eg, insulin, Byetta®, Bydureon®, or Victoza). Short-term use of insulin within this period will not be cause for exclusion if insulin was used during the treatment of an acute intercurrent illness;
* Known allergy to or serious adverse effect caused by an approved or investigational glucagon-like peptide-1 (GLP-1) receptor analog/agonist;
* Unstable cardiovascular disease;
* History of weight loss surgery or other gastrointestinal surgical procedures that could possibly interfere with the mechanism of action of GLP-1 receptor agonists;
* Based on contraindications/warnings identified with other GLP-1 receptor agonists, subjects will be excluded if they have: History, symptoms, or signs of pancreatitis or severe gastrointestinal disease (ie, gastroparesis) or Personal or family history of medullary thyroid tumors or history of Multiple Endocrine Neoplasia Syndrome Type 2;
* Clinically significant renal and/or hepatic dysfunction;
* Pregnant or lactating female subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of dose response of Glymera as measured as the change from baseline in HbA1c after 20 weeks of dosing with Glymera compared to placebo and active comparator | Baseline and 20 weeks

SECONDARY OUTCOMES:
Description of the incidence, severity, and duration of reported gastrointestinal side effects of Glymera compared to active comparator | Up to 23 weeks
Compare change from baseline in weekly fasting plasma glucose (FPG) following 20 weeks of dosing compared to placebo and active comparator | Baseline and 20 weeks
Describe the frequencies of adverse events in the treatment groups | Up to 23 weeks
Proportion of subjects reaching HbA1c targets (<7.0%) after 20 weeks of dosing | Baseline and 20 weeks

CONTACTS AND LOCATIONS:
Locations (93):
- United States (93):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Gulf Shores, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Muscle Shoals, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Goodyear, Arizona
  - Tucson, Arizona
  - Harrisburg, Arkansas
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Chula Vista, California
  - Concord, California
  - Escondido, California
  - Hawaiian Gardens, California
  - La Mesa, California
  - Los Angeles, California
  - Oceanside, California
  - San Jose, California
  - Santa Rosa, California
  - Walnut Creek, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Stamford, Connecticut
  - Brandenton, Florida
  - Brooksville, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Oviedo, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Marietta, Georgia
  - Roswell, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Council Bluffs, Iowa
  - Augusta, Kansas
  - Newton, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - New Orleans, Louisiana
  - Oxon Hill, Maryland
  - Ypsilanti, Michigan
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Fremont, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - New Windsor, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Delaware, Ohio
  - Kettering, Ohio
  - Lyndhurst, Ohio
  - Wadsworth, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Greer, South Carolina
  - Spartanburg, South Carolina
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - Hurst, Texas
  - Katy, Texas
  - Magna, Utah
  - West Jordan, Utah
  - Burke, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington
  - Kenosha, Wisconsin